CLINICAL TRIAL: NCT06979934
Title: The Effect of 3D Printing Functional Splints on Hand Function for Patients With Stroke
Brief Title: Effect of 3D Printing Functional Hand Splints for Patients With Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because the project proposal was not approved for funding, it was not carried out.
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-JIRB N202104007
Record Dates: First submitted 2021-05-23; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D printing splint group (Experimental): 3D printing splint for 8 weeks of treatment (Sixty minutes for position and twenty minutes for training a time, triple times a day)
  Interventions: Behavioral: 3D printing splint group
- functional splint group (Active Comparator): functional splint for 8 weeks of treatment (Sixty minutes for position and twenty minutes for training a time, triple times a day)
  Interventions: Behavioral: functional splint group

INTERVENTIONS:
Behavioral: 3D printing splint group — Wear 3D printing design splint for position for 60 minutes each time, plus 20 minutes of exercise which including:(1) Raise hands for 5 minutes, and bend and straighten the elbow for 5 minutes for proximal movement exercise;(2) Wear 3D printed design hand splint and change objects according to the ability of grasp, such as hold a cup, handle, eraser, pen, etc.
  Arms: 3D printing splint group
Behavioral: functional splint group — Wear functional splint for position for 60 minutes each time, plus 20 minutes of exercise which including:(1) Raise hands for 5 minutes, and bend and straighten the elbow for 5 minutes for proximal movement exercise;(2) Grasp the holder according the grasp ability, such as hold a cup, handle, eraser, pen, etc.
  Arms: functional splint group

SUMMARY:
The study is to evaluate the effect of 3D printing functional splints on hand function for patients with stroke.Twenty stroke patients with moderate motor deficits were recruited and randomized into experimental (3D printing splint) or control (functional splint) groups for 8 weeks of treatment.The performance was assessed by a blinded assessor for two times including motor, function, and feasibility.Collected data will be analyzed with nonparametric tests by SPSS version 20.0, and alpha level was set at .05.

DETAILED DESCRIPTION:
Background: Spasticity is an important factor limiting independency and activity of daily living for post-stroke patients. Splinting has been proved to be successful treatment for spasticity.3D printing technology was used to construct personalized, complicated orthosis, and one piece to reduce assembly time. The evidence most are product development, but few of study investigate the effectiveness.

Aim: To evaluate the effect of 3D printing functional splints on hand function for patients with stroke.

Methods: Twenty stroke patients with moderate motor deficits were recruited and randomized into experimental (3D printing splint) or control (functional splint) groups for 8 weeks of treatment (Sixty minutes for position and twenty minutes for training a time, triple times a day). The performance was assessed by a blinded assessor for two times included Fugl-Meyer Assessment-Upper Limb section(FMA-UE), Electromyography (EMG), Grip dynamometer, Passive Range of motion (PROM) at upper extremity, Muscle tone at upper extremity, and Disability of the arm, shoulder and hand questionnaire(DASH). The splint wearing performance and Satisfaction were recorded. Collected data will be analyzed with nonparametric tests by SPSS version 20.0, and alpha level was set at .05.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral stroke, patients with unilateral hemiplegia
* Onset is more than three months;
* Able to understand activity instructions;
* Fugl-Meyer assessment 20-50 points

Exclusion Criteria:

* Age over 75 years and under 20 years old;
* Other medical diseases that affect the execution program
* Modified Ashworth Scale of Wrist and hand greater than 2 Points
* Deformed elbow, wrist and hand joints
* Treated with botulinum toxin on the upper limbs of the affected side.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-upper extremity | Change from Baseline at 8 weeks
  The Fugl-Meyer Assessment-upper extremity (FMA-UE) measures motor impairment in the upper extremity. The assessment consists of 33 items, including movement, reflex, grasp, and coordination, and a total score of 66.The unit of measure is score.

SECONDARY OUTCOMES:
Electromyography | Change from Baseline at 8 weeks
  Record the maximum voluntary contraction (maximal voluntary contraction; MVC) of the wrist extensor muscles, total extensor muscles, and flexor muscles.The unit of measure is motor unit.
Dynanometer | Change from Baseline at 8 weeks
  The grip dynamometer was used to measure the maximum isometric strength of the hand and forearm muscles. The mean score of 3 trials was calculated. For this measurement, the elbow was placed at 90° and the forearm was placed in mid-position.The unit of measure is kilograms.
Range of motion of upper limb joints | Change from Baseline at 8 weeks
  Passive movement angle of elbow joint, wrist joint and thumb, finger metacarpophalangeal joint.The unit of measure is degree.
Disabilities of The Arm, Shoulder And Hand Questionnaire | Change from Baseline at 8 weeks
  a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. We used the subtest of Activity capacity, severity of illness.The unit of measure is score.
Side effects record | Every training session, total sessions continued to 8 weeks
  The number of side effects after intervention (such as soreness, pain, motion vertigo, injury, etc.) were recorded every day. The unit of measure is number of times.
Satisfaction questionnaire | Every training session, total sessions continued to 8 weeks
  The questionnaire is a subjective self-filling scale using a hand brace, with 5-level scores (strongly agree to strongly disagree), including aesthetics, complexity, weight, resistance, comfort, ease of wear, etc.The unit of measure is score.
Wear performance record | Every training session, total sessions continued to 8 weeks
  The wear and exercise times were recorded every day. The unit of measure is number of times.

CONTACTS AND LOCATIONS:
Overall Officials: Hsinchieh Lee, Principal Investigator — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander J, Dawson J, Langhorne P. Dynamic hand orthoses for the recovery of hand and arm function in adults after stroke: A systematic review and meta-analysis of randomised controlled trials. Top Stroke Rehabil. 2022 Mar;29(2):114-124. doi: 10.1080/10749357.2021.1878669. Epub 2021 Jan 31. PMID 33517868
- [Background] Ates, S., Haarman, C. J., & Stienen, A. H. J. A. R. (2017). SCRIPT passive orthosis: design of interactive hand and wrist exoskeleton for rehabilitation at home after stroke. 41(3), 711-723.
- [Background] Azeez, A., Gopichand, A., Shankar, N., Hanumantharao, K. J. I. J. o. E. T., & Technology. (2015). A novel prosthetic hand support for physically disabled. 29(6), 295-298
- [Background] Baronio G, Harran S, Signoroni A. A Critical Analysis of a Hand Orthosis Reverse Engineering and 3D Printing Process. Appl Bionics Biomech. 2016;2016:8347478. doi: 10.1155/2016/8347478. Epub 2016 Aug 9. PMID 27594781
- [Background] Basteris A, Nijenhuis SM, Stienen AH, Buurke JH, Prange GB, Amirabdollahian F. Training modalities in robot-mediated upper limb rehabilitation in stroke: a framework for classification based on a systematic review. J Neuroeng Rehabil. 2014 Jul 10;11:111. doi: 10.1186/1743-0003-11-111. PMID 25012864
- [Background] Cazon, A., Aizpurua, J., Paterson, A., Bibb, R., Campbell, R. I. J. V., & Prototyping, P. (2014). Customised design and manufacture of protective face masks combining a practitioner-friendly modelling approach and low-cost devices for digitising and additive manufacturing: This paper analyses the viability of replacing conventional practice with AM method to make customized protective face masks. 9(4), 251-261.
- [Background] Chang, K., Chang, J.-H., Huang, M.-W., & Lee, L.-Y. (2018). Innovative orthosis for phalanx extension neurofacilitation (iOPEN)-development of a 3D-printed hand orthosis for chronic stroke patient. Paper presented at the 2018 IEEE International Conference on Applied System Invention (ICASI).
- [Background] Chang WD, Lai PT. New design of home-based dynamic hand splint for hemiplegic hands: a preliminary study. J Phys Ther Sci. 2015 Mar;27(3):829-31. doi: 10.1589/jpts.27.829. Epub 2015 Mar 31. PMID 25931740
- [Background] Copley J, Kuipers K, Fleming J, Rassafiani M. Individualised resting hand splints for adults with acquired brain injury: a randomized, single blinded, single case design. NeuroRehabilitation. 2013;32(4):885-98. doi: 10.3233/NRE-130913. PMID 23867415
- [Background] Diment LE, Thompson MS, Bergmann JH. Three-dimensional printed upper-limb prostheses lack randomised controlled trials: A systematic review. Prosthet Orthot Int. 2018 Feb;42(1):7-13. doi: 10.1177/0309364617704803. Epub 2017 Jun 24. PMID 28649911
- [Background] Duncan PW, Propst M, Nelson SG. Reliability of the Fugl-Meyer assessment of sensorimotor recovery following cerebrovascular accident. Phys Ther. 1983 Oct;63(10):1606-10. doi: 10.1093/ptj/63.10.1606. PMID 6622535
- [Background] Emzain, Z. F., Huang, S.-C., Yang, Y.-S., & Qosim, N. J. R. M. (2020). Design and Analysis of a Dynamic Splint Based on Pulley Rotation for Post-Stroke Finger Extension Rehabilitation Device. 11(3), 477-485.
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944
- [Background] Fitzpatrick, A. P., Mohanned, M. I., Collins, P. K., & Gibson, I. J. K. E. (2017). Design of a patient specific, 3D printed arm cast. 135-142.
- [Background] Gregson JM, Leathley M, Moore AP, Sharma AK, Smith TL, Watkins CL. Reliability of the Tone Assessment Scale and the modified Ashworth scale as clinical tools for assessing poststroke spasticity. Arch Phys Med Rehabil. 1999 Sep;80(9):1013-6. doi: 10.1016/s0003-9993(99)90053-9. PMID 10489001
- [Background] Hamilton GF, McDonald C, Chenier TC. Measurement of grip strength: validity and reliability of the sphygmomanometer and jamar grip dynamometer. J Orthop Sports Phys Ther. 1992;16(5):215-9. doi: 10.2519/jospt.1992.16.5.215. PMID 18796752
- [Background] Jang SH. The recovery of walking in stroke patients: a review. Int J Rehabil Res. 2010 Dec;33(4):285-9. doi: 10.1097/MRR.0b013e32833f0500. PMID 20805757
- [Background] Katalinic OM, Harvey LA, Herbert RD, Moseley AM, Lannin NA, Schurr K. Stretch for the treatment and prevention of contractures. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD007455. doi: 10.1002/14651858.CD007455.pub2. PMID 20824861
- [Background] Liang HW, Wang HK, Yao G, Horng YS, Hou SM. Psychometric evaluation of the Taiwan version of the Disability of the Arm, Shoulder, and Hand (DASH) questionnaire. J Formos Med Assoc. 2004 Oct;103(10):773-9. PMID 15490028
- [Background] Lubbes, E. (2016). Investigation and Assessment of Upper-Limb Prosthetic Care and Business Model Design for 3D-Printed Prostheses in the Netherlands.
- [Background] Marque P, Gasq D, Castel-Lacanal E, De Boissezon X, Loubinoux I. Post-stroke hemiplegia rehabilitation: evolution of the concepts. Ann Phys Rehabil Med. 2014 Nov;57(8):520-529. doi: 10.1016/j.rehab.2014.08.004. Epub 2014 Aug 23. PMID 25282582
- [Background] Mills PB, Finlayson H, Sudol M, O'Connor R. Systematic review of adjunct therapies to improve outcomes following botulinum toxin injection for treatment of limb spasticity. Clin Rehabil. 2016 Jun;30(6):537-48. doi: 10.1177/0269215515593783. Epub 2015 Jul 21. PMID 26198891
- [Background] Munhoz, R., Moraes, C. A. d. C., Tanaka, H., & Kunkel, M. E. J. R. o. B. E. (2016). A digital approach for design and fabrication by rapid prototyping of orthosis for developmental dysplasia of the hip. 32(1), 63-73.
- [Background] Nordin N, Xie SQ, Wunsche B. Assessment of movement quality in robot- assisted upper limb rehabilitation after stroke: a review. J Neuroeng Rehabil. 2014 Sep 12;11:137. doi: 10.1186/1743-0003-11-137. PMID 25217124
- [Background] Phillips, B., Zingalis, G., Ritter, S., & Mehta, K. (2015). A review of current upper-limb prostheses for resource constrained settings. Paper presented at the 2015 IEEE global humanitarian technology conference (GHTC).
- [Background] Pizzi A, Carlucci G, Falsini C, Verdesca S, Grippo A. Application of a volar static splint in poststroke spasticity of the upper limb. Arch Phys Med Rehabil. 2005 Sep;86(9):1855-9. doi: 10.1016/j.apmr.2005.03.032. PMID 16181954
- [Background] Sakai, R., Haraguchi, M., Kanamori, M., Yamada, K., Ishida, K., & Kobayashi, Y. J. A. J. o. O. T. (2020). Development of a Finger Extension Assistance Splint for a Hemiplegic Upper Limb After Stroke-A Case Report. 16(1), 83-86.
- [Background] Santamato A, Micello MF, Panza F, Fortunato F, Picelli A, Smania N, Logroscino G, Fiore P, Ranieri M. Adhesive taping vs. daily manual muscle stretching and splinting after botulinum toxin type A injection for wrist and fingers spastic overactivity in stroke patients: a randomized controlled trial. Clin Rehabil. 2015 Jan;29(1):50-8. doi: 10.1177/0269215514537915. Epub 2014 Jun 10. PMID 24917588
- [Background] Tanabe, H., Nagao, T., & Tanemura, R. J. A. J. o. O. T. (2011). Application of constraint-induced movement therapy for people with severe chronic plegic hand. 9(1), 7-14.
- [Background] Thibaut A, Chatelle C, Ziegler E, Bruno MA, Laureys S, Gosseries O. Spasticity after stroke: physiology, assessment and treatment. Brain Inj. 2013;27(10):1093-105. doi: 10.3109/02699052.2013.804202. Epub 2013 Jul 25. PMID 23885710